CLINICAL TRIAL: NCT06651307
Title: The Effect of Neoprene Elbow Sleeves on Bench Press and Shoulder Press Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nord University (Other)
Responsible Party: Principal Investigator, Runar Jakobsen Unhjem, Associate professor, Nord University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 196225
Record Dates: First submitted 2024-10-18; First posted 2024-10-21 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-10

CONDITIONS: Healhty
Keywords: bench press; maximal strength; elbow sleeves; shoulder press; as many repetitions as possible

STUDY DESIGN:
Intervention Model Description: All subjects performed testing with and without elbow sleeves. The sequence of conditions was allocated by a randomized and counterbalanced crossover approach.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lifting with elbow sleeves (Experimental): Lifting with elbow sleeves
  Interventions: Device: Lifting with elbow sleeves
- Lifting without elbow sleeves (No Intervention): Lifting without elbow sleeves

INTERVENTIONS:
Device: Lifting with elbow sleeves — Lifting with elbow sleeves
  Arms: Lifting with elbow sleeves

SUMMARY:
We examined the effect of neoprene elbow sleeves on bench press and shoulder press perforamance in a group of healhty students.

DETAILED DESCRIPTION:
20 healhty volunteers performed one repetition maximum tests in bench press and shoulder press, with and without elbow sleeves. We also tested how many repetitions the subjects were able to lift at 85% of one repetition maximum, with and without elbow sleeves.

ELIGIBILITY:
Inclusion Criteria:

* Healthy young volunteers that participated regularly in strength training

Exclusion Criteria:

* any injuries or ailments in the upper body that restricted their ability to perform heavy bench press or shoulder press lifting

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
One repetition maximum in bench press and shoulder press | Within 2 weeks after enrollment
  One repetition maximum in bench press and shoulder press

CONTACTS AND LOCATIONS:
Locations (1):
- Nord University, Bodø, Nordland, Norway

IPD SHARING:
Plan to Share IPD: Undecided
Data is not person sensitive, and will be shared upon request.